CLINICAL TRIAL: NCT04519775
Title: HOBSCOTCH Phase III: Efficacy of Enhanced Virtual HOBSCOTCH
Brief Title: HOBSCOTCH Phase III
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Barbara Jobst, Staff Physician, Neurology, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: D12217 Phase III
Record Dates: First submitted 2020-08-17; First posted 2020-08-20 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Epilepsy
Keywords: Epilepsy Memory Problems; Self-Management
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HOBSCOTCH-V (virtual) (Experimental): Participants will receive the HOBSCOTCH intervention consisting of 1:1 sessions delivered once per week, including:
  * 1 pre-HOBSCOTCH Session (on webcam)
  * 1 educational session (on webcam)
  * 6 telephone sessions
  * 1 wrap-up session (webcam or telephone)
  Participants will also receive 3 booster sessions, via webcam or telephone, once per month.
  Interventions: Behavioral: Home Based Self-management and Cognitive Training Changes lives (HOBSCOTCH)
- Control (Other): Participants will be wait listed and will receive HOBSCOTCH-V (above) following a 6 month wait period.
  Interventions: Behavioral: Home Based Self-management and Cognitive Training Changes lives (HOBSCOTCH)

INTERVENTIONS:
Behavioral: Home Based Self-management and Cognitive Training Changes lives (HOBSCOTCH) — HOBSCOTCH is a home-based self-management program to treat cognitive symptoms and improve quality of life, while minimizing the barriers of access to care. The program is based on Problem Solving Therapy (PST) and teaches problem solving strategies and compensatory mechanisms to help manage cognitive dysfunction and enhance quality of life.
  Other Names: HOBSCOTCH

SUMMARY:
The purpose of this study is to determine the efficacy of an entirely virtual version of the home-based cognitive self-management program "HOBSCOTCH." It will test whether HOBSCOTCH can be delivered nationally from a distance utilizing e-health tools (telephone, computer, and phone).

DETAILED DESCRIPTION:
HOBSCOTCH (Home Based Self-management and Cognitive Training Changes lives) is a home-based self-management program to treat cognitive symptoms and improve quality of life, while minimizing the barriers of access to care. The program is based on Problem Solving Therapy (PST) and teaches problem solving strategies and compensatory mechanisms to help manage cognitive dysfunction and enhance quality of life.

HOBSCOTCH Phase III is a study to examine an entirely virtual version of the program. While HOBSCOTCH was shown to be effective as an in-person and telephone-based program in previous trials (HOBSCOTCH Phase I and II), this study aims to test a version of the program adapted for entirely virtual delivery. This is a single-center study, with the HOBSCOTCH intervention being delivered by staff affiliated with Dartmouth-Hitchcock Medical Center in Lebanon, NH.

ELIGIBILITY:
Inclusion Criteria:

* Age 18+
* Diagnosis of epilepsy, with controlled or uncontrolled seizures
* Subjective memory complaints
* No changes in antiepileptic and antidepressant medication regimen for 1 month, however brief discontinuation of antiepileptic medicine for inpatient video EEG evaluation is acceptable
* Literate
* Telephone access
* Internet access

Exclusion Criteria:

* Subjects self-reporting a dementing illness or a mention of a dementing illness in their medical record
* Severe mental disability or estimated IQ less than 70 per clinical judgement
* Significant visual impairment precluding reading or writing
* No reliable telephone or internet access
* No diagnosis of epilepsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2020-11-12 (Actual); Primary Completion 2024-09-26 (Actual); Study Completion 2024-11-19 (Actual)

PRIMARY OUTCOMES:
Change in quality of life | Baseline and at months 3, 6, 9, 12
  The researchers will use the Quality of Life in Epilepsy (QOLIE-31). This validated tool contains 16 multi-item scales which assess health related quality of life, emotional well-being, memory and attention deficits, medication effects, seizure control, psychosocial functioning, and health perception. Scores range from 0 to 100, with a higher score reflecting a higher quality of life.
Change in cognitive function | Baseline and at months 3, 6, 9, 12
  The researchers will use the Cognitive Function sub-scale of the NeuroQOL. This is a brief validated tool developed by the NIH for use in patients with neurological disease. Scores range from 8 to 40, with a higher score indicating better reported cognitive functioning.

SECONDARY OUTCOMES:
Change in depression | Baseline and at months 3, 6, 9, 12
  The researchers will use the Patient Health Questionnaire (PHQ-9). The PHQ-9 is a brief 9-item validated depression scale. Scores range from 0 to 27. Scores of 5, 10, 15, and 20 represent cut-offs for mild, moderate, moderately severe, and severe depression, respectively.
Change in self-management practices | Baseline and at months 3, 6, 9, 12
  The researchers will use the Adult Epilepsy Self-Management Measurement Instrument (AESMMI-65).This is a 65 item scale that assesses use of epilepsy self-management practices. Scores range from 65 to 325, with a higher score indicating more frequent use of self-management strategies.
Changes in self-reported seizure frequency | Ongoing through entire study baseline - 12 months
  The researchers will collect seizure information throughout the entire study by use of a smartphone app or paper log to track seizures daily. No range.
Changes in medication adherence | Ongoing through entire study baseline - 12 months, and at baseline and at months 3, 6, 9, 12
  Medication adherence will be collected using the Medication Adherence Rating Scale (MARS), a 10-item inventory to measure medication adherence, as well as by a daily single item medication adherence question through a smartphone app or paper log. For the MARS, scores range from 0 to 10, with a higher score indicating better adherence.
Changes in health confidence | Baseline and at months 3, 6, 9, 12
  The researchers will use the Health Confidence Score, a 4-item measure of health confidence. Scores range from 0 to 13, with a higher score indicating better health confidence.
Changes in healthcare utilization | Baseline and at months 3, 6, 9, 12
  The researchers will use the Health Care Utilization 4-item measure from the Self-Management Resource Center to capture utilization of health services in the last 6 months. No range.
Changes in overall well-being | Ongoing through entire study baseline - 12 months
  The researchers will collect daily well-being information throughout the entire study by use of a smartphone app or paper log and a basic single item Likert-scale of well-being. No range.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Jobst, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center and Dartmouth College
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Caller TA, Secore KL, Ferguson RJ, Roth RM, Alexandre FP, Henegan PL, Harrington JJ, Jobst BC. Design and feasibility of a memory intervention with focus on self-management for cognitive impairment in epilepsy. Epilepsy Behav. 2015 Mar;44:192-4. doi: 10.1016/j.yebeh.2014.12.036. Epub 2015 Feb 27. PMID 25731132
- [Background] Caller TA, Ferguson RJ, Roth RM, Secore KL, Alexandre FP, Zhao W, Tosteson TD, Henegan PL, Birney K, Jobst BC. A cognitive behavioral intervention (HOBSCOTCH) improves quality of life and attention in epilepsy. Epilepsy Behav. 2016 Apr;57(Pt A):111-117. doi: 10.1016/j.yebeh.2016.01.024. Epub 2016 Mar 2. PMID 26943948